CLINICAL TRIAL: NCT03259919
Title: Metformin Treatment of Pregnant Women With Polycystic Ovary Syndrome: a Pilot Study
Acronym: pilPregMet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 220800
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Metformin; Pregnancy outcome; Androgens
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin 850 mg x 2 daily
  Interventions: Drug: Metformin
- placebo (Placebo Comparator): Placebo 1 tablet x 2 daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg x 1 per day for the first week, and 850 mg x 2 per day for the rest of the study period.. Orally. From inclusion (before gestational week 8) to delivery. Verbal and written diet and lifestyle advices at inclusion to the study. In addition 1 mg tablet of folate and one daily multivitamin tablet.
  Other Names: metformin from Weifa 425 mg / tablet
  Arms: Metformin
Drug: Placebo — Placebo, 2 tablets x 1 daily for the first week, and 2 tablets x 2 for the rest of the study period.Orally. From inclusion (that is before gestational week 12) to delivery. Verbal and written diet and lifestyle advices at inclusion to the study. In addition 1 mg tablet of folate and one daily multivitamin tablet.
  Other Names: Placebo from Weifa
  Arms: placebo

SUMMARY:
To investigate the effect of metformin on pregnancy complications and pregnancy outcome in the II. and III. trimester of pregnancy in women with polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis polycystic ovary syndrome (PCOS ) before pregnancy
* BMI 27-40 kg/m2
* Human chorionic gonadotropin, beta subunit (HCG-beta) verified pregnancy week 5-8
* At least one of the following criteria: (1) serum testosteron > 2,5 nmol/L; (2) Sex hormone binding globulin (SHBG) < 30 nmol; (3) Fasting C-peptid > 1,0 nmol/L; (4) Menstrual disturbances: oligo-/amenorrhea or metrorrhagia; (5) Hirsutism

Exclusion Criteria:

* known liver disease or ALAT > 60 IU/L
* S-creatinin > 130 micromol/L
* diabetes mellitus
* alcohol or drug abuse
* peroral steroid treatment (except inhalation steroids)
* use of cimetidine, anticoagulant, erythromycin or other macrolides
* not suitable for other reasons

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2000-10 (Actual); Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Dehydroepiandrosterone sulfate (DHEAS) | up to delivery
  (µmol/l) Analysed in serum, from venous blood samples from the mother and venous and arterial umbilical cord blood (separately) collected within 1 h of birth. Measured using a competitive immunoassay on an Immulite 2000 analyser using the reagents and calibrators supplied by the manufacturer (Diagnostic Products Corp., USA)
Androstenedione | up to delivery
  Analysed in serum, from venous blood samples from the mother and venous and arterial umbilical cord blood (separately) collected within 1 h of birth. measured by a double antibody technique on an Elecsys 2010 analyser (Roche Diagnostics GmbH, Germany) using reagents and calibrators supplied by the manufacturer
Testosterone | up to delivery
  Analysed in serum, from venous blood samples from the mother and venous and arterial umbilical cord blood (separately) collected within 1 h of birth. measured by a double antibody technique on an Elecsys 2010 analyser (Roche Diagnostics GmbH, Germany) using reagents and calibrators supplied by the manufacturer
Sex hormone binding globulin (SHBG) | up to delivery
  (nmol/l) Analysed in serum, from venous blood samples from the mother and venous and arterial umbilical cord blood (separately) collected within 1 h of birth. Measured using a competitive immunoassay on an Immulite 2000 analyser using the reagents and calibrators supplied by the manufacturer (Diagnostic Products Corp., USA)
Free testosterone index | up to delivery
  Calculated as total testosterone divided by SHBG and multiplied by a factor of 100. SHBG measured using a competitive immunoassay on an Immulite 2000 analyser using the reagents and calibrators supplied by the manufacturer (Diagnostic Products Corp., USA)

SECONDARY OUTCOMES:
Occurence of pregnancy complications | up to 6 weeks post partum
  Gestational diabetes (GDM) defined according to World Health Organization (1998) criteria, i.e. 2 h plasma glucose values ≥7.8 mmol/l during an Oral Glucose Tolerance Test (OGTT) with 75 g. Uncomplicated GDM treated with dietary advice only was not ranked among the complications in this study. Pre-eclampsia defined as a blood pressure ≥140/90mmHg with concomitant albuminuria ≥0.3 g/24 h measured on two separate occasions after gestational week 20. Premature delivery was defined as delivery before gestational week 37 + 0 according to an estimated date of delivery, based on mid-trimester ultrasound scan
Pregnancy outcome - gestational age | after delivery
  Gestational age at birth (days)
Pregnancy outcome - gestational length | after delivery
  Gestational length (cm) measured at birth
Pregnancy outcome - head circumference | after delivery
  Head circumference (cm) measured at birth.
Pregnancy outcome - birthweight | after delivery
  Birthweight (g) measured at birth
Pregnancy outcome - placental weight | after delivery
  Placental weight (g) measured at birth
Pregnancy outcome - Agpar score at 5 minutes | after delivery
  Apgar score at 5 minutes
Pregnancy outcome - Agpar score at 10 minutes | after delivery
  Apgar score at 10 minutes
Pregnancy outcome - umbilical artery pH | after delivery
  Umbilical artery pH measured in umbilical artery blood, immediately after delivery on a Rapidlab 248pH/Blood Gas Analyzer, using reagents and calibrators supplied by the manufacturer (Bayer Corp., USA)

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Departments of Obstetrics and Gynecology and Endocrinology, St. Olav's Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vanky E, Salvesen KA, Heimstad R, Fougner KJ, Romundstad P, Carlsen SM. Metformin reduces pregnancy complications without affecting androgen levels in pregnant polycystic ovary syndrome women: results of a randomized study. Hum Reprod. 2004 Aug;19(8):1734-40. doi: 10.1093/humrep/deh347. Epub 2004 Jun 3. PMID 15178665
- [Result] Hanem LGE, Stridsklev S, Juliusson PB, Salvesen O, Roelants M, Carlsen SM, Odegard R, Vanky E. Metformin Use in PCOS Pregnancies Increases the Risk of Offspring Overweight at 4 Years of Age: Follow-Up of Two RCTs. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1612-1621. doi: 10.1210/jc.2017-02419. PMID 29490031
- [Derived] Ryssdal M, Skage JE, Jarmund AH, Hanem LGE, Lovvik TS, Giskeodegard GF, Iversen AC, Vanky E. Metformin Treatment in PCOS Pregnancies Reduces Maternal Infections and Increases the Risk of Allergies and Eczema in the Offspring: Post Hoc Analyses of Two Randomised Controlled Trials and One Follow-Up Study. BJOG. 2025 Nov;132(12):1823-1832. doi: 10.1111/1471-0528.18320. Epub 2025 Aug 11. PMID 40785326
- [Derived] Nordtvedt E, Kessler J, Ebbing C, Acharya G, Lovvik TS, Salvesen KA, Salvesen O, Vanky E, Kahrs BH. Placental and cerebral circulation in fetuses of mothers with polycystic ovary syndrome and the effect of Metformin exposure. BMC Pregnancy Childbirth. 2025 Jul 10;25(1):749. doi: 10.1186/s12884-025-07866-9. PMID 40640743
- [Derived] Ujvari D, Trouva A, Hirschberg AL, Vanky E. Maternal serum levels of prokineticin-1 related to pregnancy complications and metformin use in women with polycystic ovary syndrome: a post hoc analysis of two prospective, randomised, placebo-controlled trials. BMJ Open. 2023 Nov 21;13(11):e073619. doi: 10.1136/bmjopen-2023-073619. PMID 37989369
- [Derived] Trouva A, Alvarsson M, Calissendorff J, Asvold BO, Vanky E, Hirschberg AL. Thyroid Status During Pregnancy in Women With Polycystic Ovary Syndrome and the Effect of Metformin. Front Endocrinol (Lausanne). 2022 Feb 21;13:772801. doi: 10.3389/fendo.2022.772801. eCollection 2022. PMID 35265033
- [Derived] Underdal MO, Salvesen O, Henriksen AH, Andersen M, Vanky E. Impaired Respiratory Function in Women With PCOS Compared With Matched Controls From a Population-Based Study. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz053. doi: 10.1210/clinem/dgz053. PMID 31613965
- [Derived] Underdal MO, Stridsklev S, Oppen IH, Hogetveit K, Andersen MS, Vanky E. Does Metformin Treatment During Pregnancy Modify the Future Metabolic Profile in Women With PCOS? J Clin Endocrinol Metab. 2018 Jun 1;103(6):2408-2413. doi: 10.1210/jc.2018-00485. PMID 29659896